CLINICAL TRIAL: NCT00496509
Title: A Phase I, Open-Label Study To Assess The Effect of ZD6474 (ZACTIMA) On Vascular Permeability In Patients With Advanced Colorectal Cancer and Liver Metastases
Brief Title: Phase I Efficacy On Vascular Permeability In Patients With Advanced Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D4200C00050
Record Dates: First submitted 2007-07-03; First posted 2007-07-04 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Colorectal Cancer
Keywords: ZD6474; Colorectal Cancer; Liver Metastases; Biomarkers
MeSH Terms: conditions — Colorectal Neoplasms | interventions — vandetanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ZD6474 (vandetanib) 100mg (Experimental)
  Interventions: Drug: ZD6474 (Zactima) 100mg; Procedure: Dynamic Contrast-Enhanced Magnetic Resonance Imaging (DCE-MR); Procedure: Biomarker Draws
- ZD6474 (vandetanib) 300mg (Experimental)
  Interventions: Procedure: Dynamic Contrast-Enhanced Magnetic Resonance Imaging (DCE-MR); Procedure: Biomarker Draws; Drug: ZD6474 (Zactima) 300mg

INTERVENTIONS:
Drug: ZD6474 (Zactima) 100mg
  Arms: ZD6474 (vandetanib) 100mg
Procedure: Dynamic Contrast-Enhanced Magnetic Resonance Imaging (DCE-MR)
Procedure: Biomarker Draws
Drug: ZD6474 (Zactima) 300mg
  Arms: ZD6474 (vandetanib) 300mg

SUMMARY:
A Phase I, Open-Label Study To Assess The Effect of ZD6474 (ZACTIMA) On Vascular Permeability In Patients with Advanced Colorectal Cancer and Liver Metastases.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic colorectal adenocarcinoma (stage IV) with at least 1 measurable hepatic lesion of 20 mm or more on MRI and for whom no standard therapy is available.
* WHO Performance status 0 - 2.
* Life expectancy of at least 12 weeks

Exclusion Criteria:

* Brain metastases or spinal cord compression, unless treated at least 4 weeks before entry and stable without steroid treatment for 10 days or greater.
* Last dose of prior chemotherapy must be discontinued at least 4 weeks before the start of study treatment.
* Last dose of radiotherapy received within 4 weeks before the start of study treatment excluding palliative radiotherapy.
* Prior treatment with VEGFR TKIs
* Serum bilirubin . 1.5 x the upper limit of reference range.
* Serum creatinine >1.5 x ULRR or Creatinine clearance (as determined by the Cockcroft - Gault method) less than or equal to 50 mL/min.
* ALT or AST >5 x ULRR
* ALP >5 x ULRR
* Evidence of severe or uncontrolled systemic disease or any concurrent conditions which in the investigators opinion make it undesirable for the patient to participate in the study or would jeopardize compliance with the protocol.
* Any unresolved toxicity greater than CTCAE Grade 2 for previous anti-cancer therapy.
* Significant cardiovascular event within 3 months before entry, or presence of cardiac disease that in the opinion of the investigator increases the risk of ventricular arrhythmia.
* History of arrhythmia which is symptomatic or requires treatment (CTCAE grade 3) or asymptomatic sustained ventricular tachycardia. Atrial fibrillation, controlled by medication is not excluded.
* Congenital long QT syndrome or 1st degree relative with sudden unexplained death under of 40 years of age.
* Presence of Left Bundle Branch Block.
* QTc with Bazett's correction unmeasurable or greater than or equal to 480 msec or greater of screening ECG.
* Potassium <4.0 mmol/L despite supplementation, serum calcium (ionized or adjusted for albumin), or magnesium out of normal range despite supplementation.
* Women who are pregnant or breast feeding.
* Any concomitant medications that may cause QTc prolongation or induce or induce Torsades de Pointes or induce CTP3A4 function.
* Hypotension not controlled by medical therapy.
* Participation in a clinical study of any investigational pharmaceutical agent within 30 days prior to commencing study treatment.
* Major surgery within 4 weeks or incompletely healed surgical incision.
* Previous or current malignancies of other histologies within the last 5 years, with the exception of in situ carcinoma of the cervix and adequately treated basal cell or Squamous cell carcinoma of the skin.
* Any contraindications to MRI scans.
* Involvement in the planning or conduct of the study.
* Previous enrollment or randomization of treatment in the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-08; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Assess by dynamic contrast-enhanced magnetic resonance imaging the effect of once daily dosing with ZD6474 on tumour perfusion and vascular permeability in patients with advanced colorectal cancer and liver metastases. | Up to 57 days.

SECONDARY OUTCOMES:
Assessment of appropriate Pharmacokinetic parameters | Predetermined timepoints after dose administration
  The exposure to ZD6474 in patients with advanced colorectal cancer and liver metastases by assessment of: maximum plasma concentration after single and at steady state (C max and Css, max); time to reach C max and Css, max (tmax); minimum plasma concentration before and at steady state (Cmin and Css, min); area under plasma concentration-time curve from zero to 24 h and at steady state (AUC(0-24) and AUCss); total body clearance of drug from plasma after an oral dose (CL/F): accumulation ratio (Rac) and fraction of ZD6474 unbound (fu).
Determine the population PK of ZD6474 and assess the relationship between both free and total plasma PK and measures of Pharmacological activity | Predetermined timepoints after dose administration
  Determination of the population PK of ZD6474 and the assessment of the relationship between both free and total plasma PK and measures of pharmacological activity by assessment of individual predicted plasma concentrations, individual predicted CL/F, AUCss, Css, max, and AUC to the point up to the scan.
Assessment of the effectiveness of ZD6474 as measured by objective response rate and progression free survival based on RECIST. | Every 8 weeks during the study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Principal Investigator — Sanofi
Locations (1):
- Research Site, Freiberg, Germany

REFERENCES:
- [Background] Mross K, Fasol U, Frost A, Benkelmann R, Kuhlmann J, Buchert M, Unger C, Blum H, Hennig J, Milenkova TP, Tessier J, Krebs AD, Ryan AJ, Fischer R. DCE-MRI assessment of the effect of vandetanib on tumor vasculature in patients with advanced colorectal cancer and liver metastases: a randomized phase I study. J Angiogenes Res. 2009 Sep 21;1:5. doi: 10.1186/2040-2384-1-5. PMID 19946413